CLINICAL TRIAL: NCT07195396
Title: A Randomized, Double-blind, Moncentric, Cross-over Study to Collect Human Serum After Ingestion of Hydrolyzed Collagen Peptides.
Brief Title: To Collect Enriched Human Serum Following Hydrolyzed Collagen Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BTS2215/25
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Women
Keywords: collagen peptides; collagen hydrolysates; enriched human serum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Collagen hydrolysate 1 (Active Comparator): 10g single oral dose dissolved in water
  Interventions: Dietary Supplement: Collagen hydrolysate 1
- Collagen hydrolysate 2 (Active Comparator): 10g single oral dose dissolved in water
  Interventions: Dietary Supplement: Collagen hydrolysate 2
- Collagen hydrolysate 3 (Active Comparator): 10g single oral dose dissolved in water
  Interventions: Dietary Supplement: Collagen hydrolysate 3
- Collagen hydrolysate 4 (Active Comparator): 10g single oral dose dissolved in water
  Interventions: Dietary Supplement: Collagen hydrolysate 4
- Collagen hydrolysate 5 (Active Comparator): 10g single oral dose dissolved in water
  Interventions: Dietary Supplement: Collagen hydrolysate 5

INTERVENTIONS:
Dietary Supplement: Collagen hydrolysate 1 — 10g single oral dose dissolved in water
  Other Names: Collagen peptides
  Arms: Collagen hydrolysate 1
Dietary Supplement: Collagen hydrolysate 2 — 10g single oral dose dissolved in water
  Other Names: collagen peptides
  Arms: Collagen hydrolysate 2
Dietary Supplement: Collagen hydrolysate 3 — 10g single oral dose dissolved in water
  Other Names: collagen peptides
  Arms: Collagen hydrolysate 3
Dietary Supplement: Collagen hydrolysate 4 — 10g single oral dose dissolved in water
  Other Names: collagen peptides
  Arms: Collagen hydrolysate 4
Dietary Supplement: Collagen hydrolysate 5 — 10g single oral dose dissolved in water
  Other Names: collagen peptides
  Arms: Collagen hydrolysate 5

SUMMARY:
This randomized, double-blind, monocentric, five-way cross-over study aims to collect human serum and plasma samples at 1 and 2 hours after ingestion of hydrolyzed collagen peptides. The enriched sera will be used for ex vivo/ in vitro experiments on skin keratinocytes, fibroblasts, and other cell types to explore the beneficial effects of bioactive collagen peptides. Blood will also be analyzed for amino acid profiles and collagen-derived peptides.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able and willing to sign the Informed Consent Form prior to screening evaluations
* Age: 35 - 45 years
* Women
* BMI: 19 - 25 kg/m2
* Non-smoker
* Participant is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry and haematology at screening

Exclusion Criteria:

* Relevant history or presence of any severe medical disorder, potentially interfering with this study (e.g. mal absorption, chronic gastro-intestinal diseases, heavy depression, diabetes, significant CVD events, acute cancers within last 3 years except basal cell carcinoma of the skin, etc.)
* Significant changes in lifestyle or medication (within last 3 mo.) or surgical intervention or surgical procedure such as bariatric surgery
* Application of corticoids (intravenously, orally or intraarticularly) and other immune-suppressing drug (within last 2 weeks)
* Blood donation within 1 month prior to study start or during study
* Low haemoglobin levels < 12 g/dL
* Regular intake of drugs or supplements possibly interfering with this study within 2 weeks prior to study start or during study (stable medication since > 3 months e.g. L-Thyroxin, blood pressure medication etc. allowed)
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid, anticoagulants (e.g. Marcumar), diuretics, thiazides), which in the investigator's opinion would impact participant safety
* Not willing to avoid intake of pain relievers e.g. Paracetamol or Ibuprofen 24h prior to study days
* Participants with history of drug, alcohol or other substance abuse, or other factors limiting their ability to co-operate during the study
* History of hypersensitivity to fish
* HIV-infection, acute or chronic hepatitis B and C infection
* Known pregnancy, breast feeding or intention to become pregnant during the study. A pregnancy test will be conducted during screening and visits 1-5.
* Participation in another clinical study within the last 4 weeks and concurrent participation in another clinical study
* Anticipating any planned changes in lifestyle for the duration of the study
* Participants considered inappropriate for the study by investigators, including participants who are unable or unwilling to show compliance with the protocol

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2025-10-22 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
collagen-derived di- and tripeptides | 0-120 minutes
  Change from baseline in serum concentration of collagen-derived di- and tripeptides (e.g., Pro-Hyp, Hyp-Gly in nanogram/mL) at 1 hour and 2 hours post-intake, measured by LC-MS/MS

SECONDARY OUTCOMES:
Amino acids profile | 0-120 minutes
  Change from baseline in plasma amino acid profile (e.g., hydroxyproline, proline, glycine in microgram/mL) at 1 hour and 2 hours post-intake, measured by LC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Praneeth Reddy Kuninty, PhD, Principal Investigator — Rousselot BV
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No